CLINICAL TRIAL: NCT01671943
Title: Evaluation of Safety and Feasibility of ICE-SENSE3TM , a Cryotherapy Device for Office-based Ultrasound- Guided Treatment of Breast Cancer
Brief Title: Cryotherapy for Breast Cancer Trial
Acronym: ICE-BREACCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IceCure Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICMBC-01
Record Dates: First submitted 2012-06-27; First posted 2012-08-24 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Breast Carcinoma
Keywords: small malignant invasive breast tumors
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breast carcinoma up to 2.0 cm (Experimental)
  Interventions: Device: Ice-Sense3TM

INTERVENTIONS:
Device: Ice-Sense3TM — Ice-Sense Cryoprobe

SUMMARY:
The purpose of this study is to evaluate the clinical feasibility and safety of the ICESENSE3TM cryotherapy system for the ablation of small malignant invasive breast tumors.

ELIGIBILITY:
Inclusion Criteria:

* Unifocal primary invasive ductal breast carcinoma diagnosed by core needle biopsy. Patients with contralateral disease will remain eligible. Note: Results of ER, PR, HER-2/neu must be obtained on pre-registration needle core biopsy material.
* Tumor size ≤ 2.0 cm in greatest diameter as measured by breast ultrasound, MRI and mammogram. The largest dimension measured will be used to determine eligibility.
* Tumor enhancement on MRI
* Tumor with <25% intraductal components in the aggregate.
* Non-pregnant and non-lactating patients. Patients of childbearing potential must have a negative serum or urine pregnancy test. NOTE: Peri-menopausal women must be amenorrheic for > 12 months to be considered not of childbearing potential.
* Adequate breast size for safe cryoablation. Patients with breasts too small to allow safe cryoablation are not eligible as the minimal thickness of the breast tissue does not lend itself to cryoablation. NOTE: The minimal distance of tumor margins from the breast skin should be analogous to the surgical margins of a lumpectomy.

Exclusion Criteria:

* Patients with multifocal and/or multicentric ipsilateral breast cancer, multifocal calcifications, or evidence of excessive DCIS.
* History of rotational vacuum assisted core biopsies, en bloc open surgical biopsy and/or lumpectomy for diagnosis/treatment of the index breast cancer.
* Prior or planned neoadjuvant chemotherapy for breast cancer.
* Patients with thrombocytopenia and or any other coagulation abnormality

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The rate of complete tumor ablation in patients treated with cryoablation, with complete tumor ablation defined as no remaining invasive or in-situ carcinoma present upon pathological examination of the surgical resection specimen | One month

SECONDARY OUTCOMES:
Adverse events | One month
  To describe the adverse events associated with cryoablation in these patients.
Pain assessment | One month
  To prospectively gather pain assessment data before and after cryoablation and after surgical resection in these patients

CONTACTS AND LOCATIONS:
Overall Officials: David Pavlista, MD, Principal Investigator
Locations (1):
- Oncogynecological Center, Department of Obstetrics and Gynecology, First Faculty of Medicine, Charles University in Prague and General University Hospital in Prague Prague, Czech Republic, Prague, Czechia